CLINICAL TRIAL: NCT04283591
Title: The Effectiveness of Acupuncture Treatment for Post-Stroke Depression and Anxiety Disorder: Prospective, Randomized, Controlled Trial
Brief Title: The Effectiveness of Acupuncture Treatment for Post-Stroke Depression and Anxiety Disorder.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstPRMTRH-PSD
Record Dates: First submitted 2020-02-22; First posted 2020-02-25 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Post-stroke Depression; Anxiety Disorders
Keywords: stroke; acupuncture; depression; anxiety
MeSH Terms: conditions — Anxiety Disorders; Stroke; Depression | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Intervention (Experimental): Acupuncture Treatment Group: will get acupuncture treatment which will be applied to Baihui (DU20), Yintang (EX-HN3) points and bilateral Tai Chong (LR3), Hegu (LI4) points for 4 weeks, twice a week. They also will continue to receive the conventional rehabilitation programme.
  Interventions: Procedure: Acupuncture Treatment; Other: Conventional Rehabilitation Programme
- No Intervention (Other): Control Group: will be included in the conventional rehabilitation programme and no interventional procedures will be made.
  Interventions: Other: Conventional Rehabilitation Programme

INTERVENTIONS:
Procedure: Acupuncture Treatment — Acupuncture Treatment Group will get acupuncture treatment which will be applied to Baihui (DU20), Yintang (EX-HN3) points of the hemiplegic side and bilateral Tai Chong (LR3), Hegu (LI4) points for 4 weeks, twice a week.
  Arms: Experimental Intervention
Other: Conventional Rehabilitation Programme — They will continue to receive the conventional rehabilitation programme.

SUMMARY:
Poststroke depression is seen with a frequency of up to 30%. Drug options for depression and accompanying sleep problems are limited; In addition, effective doses cannot be increased depending on the comorbidities of the patients and the side effect profiles and drug interactions of the drugs used. Acupuncture has been used in Chinese traditional medicine for more than 2000 years and there are findings that it has positive effects in post-stroke depression and anxiety disorders.

The aim of this study is to examine the effectiveness and reliability of acupuncture treatment in depression and anxiety disorders developing after stroke and to reduce the need for multiple drugs and / or high-dose medication in the treatment of these complications.

The hypothesis of the study: Acupuncture is an effective and reliable treatment method for depression and anxiety disorders in stroke patients.

DETAILED DESCRIPTION:
Patients who receive inpatient stroke rehabilitation at Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Physical Medicine and Rehabilitation Clinic, will be included in the study by the inclusion and exclusion criteria. Their informed consent will be received. Initially, clinical and demographic data of all patients will be noted. Participants who volunteered for the study will be separated into the acupuncture treatment group and the control group by simple random sampling. Both the acupuncture treatment group and the control group will be included in the conventional rehabilitation program 2 hours a day, 7 days a week, for 8 weeks. In addition the acupuncture treatment group will get acupuncture treatment which will be applied to Baihui (DU20), Yintang (EX-HN3) points and bilateral Tai Chong (LR3), Hegu (LI4) points for 4 weeks, twice a week. During the application, the feeling of De Qi will be taken and the application will take 20 minutes. Measurements; Hamilton Depression Rating Scales, Hamilton Anxiety Rating Scales, Pittsburg Sleep Quality Index, Barthel Index, and change in psychiatric drug use will be assessed at baseline (week 0), 4th and 8th week post-treatment. The adverse events observed during the study will be noted and the compliance of patients in each application will be questioned by visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 2 months maximum 6 months after stroke
* Volunteering for study
* Mini-Mental State Examination >17
* Patients with Hamilton Depression Rating Scale> 7 and/or Hamilton Anxiety Rating Scale> 4 assessed by the psychiatrist

Exclusion Criteria:

* Insomnia and depression before a stroke
* Aphasic patients
* Sleep Apnea Syndrome
* Psychiatric Disorders (Learning disabilities, Mental disorder, Autism)
* Decompensated cardiac, kidney, hepatic failure
* Infection on Acupuncture Points
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | 1 month
  Assessed on 17 definitions, regarding the status of patient with a scale between 0 to 4.
Hamilton Anxiety Rating Scale | 1 month
  Assessed on 14 definitions, regarding the status of patient with a scale between 0 to 4.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | 1 month
  Assessed on 11 definitions, regarding the status of patient with a scale between 0 to 3.
Barthel Index | 1 month
  Assessed on 10 definitions, regarding the status of patient with a scale between 0 to 15.
Up-to-date Psychiatric Drug Use | 1 month
  Any change on previous drug dose or any newly prescribed drug will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Eser Kalaoğlu, MD, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Paolucci S. Epidemiology and treatment of post-stroke depression. Neuropsychiatr Dis Treat. 2008 Feb;4(1):145-54. doi: 10.2147/ndt.s2017. PMID 18728805
- [Background] Zhang ZJ, Chen HY, Yip KC, Ng R, Wong VT. The effectiveness and safety of acupuncture therapy in depressive disorders: systematic review and meta-analysis. J Affect Disord. 2010 Jul;124(1-2):9-21. doi: 10.1016/j.jad.2009.07.005. Epub 2009 Jul 26. PMID 19632725
- [Background] Li M, Zhang B, Meng Z, Sha T, Han Y, Zhao H, Zhang C. Effect of Tiaoshen Kaiqiao acupuncture in the treatment of ischemic post-stroke depression: a randomized controlled trial. J Tradit Chin Med. 2017 Apr;37(2):171-8. doi: 10.1016/s0254-6272(17)30041-9. PMID 29960288
- [Derived] Kalaoglu E, Kesiktas FN, Bucak OF, Atasoy M, Gunderci A. Effectiveness of acupuncture treatment in post-stroke depression and anxiety disorders: a prospective, randomized, controlled, single-blind study. Acupunct Med. 2024 Dec;42(6):319-325. doi: 10.1177/09645284241298294. Epub 2024 Nov 26. PMID 39587915